CLINICAL TRIAL: NCT06832410
Title: A Phase 3 Study to Evaluate the Efficacy, Safety, and Tolerability of VX-880 in Subjects With Type 1 Diabetes With a Kidney Transplant
Brief Title: An Efficacy, Safety, and Tolerability Study of VX-880 in Participants With Type 1 Diabetes With a Kidney Transplant
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX23-880-102
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes; Kidney Transplant
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Biological Products; Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VX-880 (Experimental)
  Interventions: Biological: Biological/Vaccine

INTERVENTIONS:
Biological: Biological/Vaccine — Infused into the hepatic portal vein.
  Other Names: Zimislecel; Formerly known as STx-02

SUMMARY:
This study will evaluate the efficacy, safety, and tolerability of VX-880 in participants with Type 1 Diabetes (TID) with a kidney transplant.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical history of T1D with greater than or equal to (≥)5 years of insulin dependence
* Taking a stable immunosuppression regimen of tacrolimus and mycophenolate mofetil, mycophenolate sodium, or sirolimus for at least 4 weeks
* Consistent use of continuous glucose monitor (CGM) for at least 4 weeks before Screening and willingness to use CGM for the duration of the study

Key Exclusion Criteria:

* Prior islet cell transplant, organ transplant (other than kidney transplant), or cell therapy, except prior pancreatic graft that failed within the first 4 weeks
* Participants had >1 kidney transplant procedure

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-09-17 (Estimated); Study Completion 2027-09-17 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants who are Insulin Independent | At 1 year After VX-880 infusion

SECONDARY OUTCOMES:
Proportion of participants who achieve insulin independence and are insulin independent 12 months later | 1 year after achieving insulin independence
Change from Baseline in glycosylated hemoglobin (HbA1c) | Baseline, At 1 year After VX-880 infusion
Proportion of Participants who Maintain Insulin Independence for at least 1 year | From VX-880 infusion to End of Study (up to 2 years)
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Signing of informed consent to End of Study (up to 2 years)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (3):
  - Perelman Center for Advanced Medicine - Endocrinology, Philadelphia, Pennsylvania
  - Montefiore Clinical and Translational Research Center - Endocrinology, Pittsburgh, Pennsylvania
  - UW University Hospital - Endocrinology, Madison, Wisconsin
- Canada (2):
  - Toronto General Hospital - Endocrinology, Toronto
  - Vancouver General Hospital - Gordon and Leslie Diamond Health Care Centre, Vancouver
- Saudi Arabia (2):
  - King Abdullah International Medical Research Center (KAIMRC) - Riyadh - Endocrinology, Riyadh
  - King Faisal Specialist Hospital & Research Centre - Riyadh - Endocrinology, Riyadh

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing